CLINICAL TRIAL: NCT05528159
Title: Perioperative Lung Ultrasound Score (LUS) Changes in Robotic and Laparoscopic Urologic Surgeries: A Prospective Observational Trial
Brief Title: Lung Ultrasound Score (LUS) Change in Robotic and Laparoscopic Urologic Surgeries
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meltem Savran Karadeniz, Associate Professor, Istanbul University
Other Study IDs: 2022/1056
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Robotic and Laparoscopic Urologic Surgery Group: Patients scheduled for robotic/laparoscopic urologic surgeries that will be performed under supine and trendelenburg position
  Interventions: Procedure: Intraabdominal CO2 insufllation

INTERVENTIONS:
Procedure: Intraabdominal CO2 insufllation — Patients will receive intraabdominal CO2 insufflation and will be operated under trendelenburg position

SUMMARY:
Robotic and laparoscopic surgeries are tend to cause lung atelectasis due to the insufflation of CO2 into abdomen. However, ultrasonographic measurement for this phenomenon and its clinical use is not well investigated. In this particular study, It is aimed to observe lung ultrasound score (LUS) changes in robotic and laparoscopic supine position surgeries such as prostatectomies and cystectomies. LUS is a pragmatic measurement method that calculates the degree of atelectasis and consolidation in the lungs. Both hemithoraxes are separated into 3 different segments with vertical lines (one between the parasternal line and anterior axillary line, one between the anterior and posterior axillary line, and one posterior to the posterior axillary line). These vertical segments are also divided into two with an horizontal line on the nipple. Lung ultrasonography is applied in all 12 zones for both lungs in the intercostal regions and a scoring system is used. Accordingly, pure A lines (transverse frequent lines) reflects normal lung tissue with no consolidation and scored as zero points (Also named "A"). If less than 4 B lines (vertical lines reflecting some degree of consolidation) is observed, it refers to 1 point (named "B1"). 4 or more B lines refers to 2 points (B2), and if wide and coalesced B lines or patchy pleural line is observed that refers to 3 points (C). All evaluations will be made in supine position.

In this trial, LUS will be applied in three different time points:

T1: 5 minutes after orotracheal intubation T2: At the end of surgery, before extubation (under deep anesthetic state) T3: 30 minutes after extubation, in postanesthesia care unit During the surgery and the postoperative care period standart monitorization and mechanical ventilation data will be gathered. Also intraoperative and postoperative blood gas analysis will be obtained to observe oxygenation changes.

This study is planned as a prospective observational study and our hypothesis is that LUS scores would be lower in acute postoperative period with robotic and laparoscopic surgeries. Therefore primary outcome is the numeric change in T3 and T1. Secondarily, LUS scores will be evaluated between robotic group and laparoscopic group patients for all time points.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Laparoscopic urologic surgeries
* Robotic urologic surgeries
* Surgeries under supine and trendelenburg position

Exclusion Criteria:

* Known lung disease
* Emergency surgeries
* Known cardiac failure
* Known pulmonary hypertension
* Patients receiving inhaled agents
* Patients requiring lateral position surgeries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for semi-elective/elective robotic and laparoscopic urologic surgeries that require supine/trendelenburg
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
LUS change between T3 and T1 | Up to 6 hours
  LUS will be evaluated at the start of the surgery right after intubation (T1) and 30 minutes after the extubation (T3). LUS refers to "lung ultrasound score" . Accordingly, one hemithorax is divided into 6 zones where the ultrasound probe is placed. If there is only A lines (no consolidation) observed, it is accepted as zero points. If there are three or less B lines (vertical lines that move with the respiration), it refers to 1 point. Four or more vertical B lines refer to 2 points, and lastly distinct visible atelectasis with converged B lines and disrupted pleura refer to 3 points. In total, ultrasonography is applied on 12 different zones, and sum of the points show the actual LUS. Less points mean lungs with better condition, and higher points reflect lungs with atelectasis and consolidation. Therefore a 36 points LUS indicates severely injured lungs.

SECONDARY OUTCOMES:
Delta T (T2-T1) and surgical duration relation | Up to 6 hours
  Intraoperative LUS change will be evaluated in relation to surgical duration. LUS refers to "lung ultrasound score" . Accordingly, one hemithorax is divided into 6 zones where the ultrasound probe is placed. If there is only A lines (no consolidation) observed, it is accepted as zero points. If there are three or less B lines (vertical lines that move with the respiration), it refers to 1 point. Four or more vertical B lines refer to 2 points, and lastly distinct visible atelectasis with converged B lines and disrupted pleura refer to 3 points. In total, ultrasonography is applied on 12 different zones, and sum of the points show the actual LUS. Less points mean lungs with better condition, and higher points reflect lungs with atelectasis and consolidation. Therefore a 36 points LUS indicates severely injured lungs.
Perioperative PaO2 analysis and its relation to T3 LUS | Up to 6 hours
  PaO2 values will be evaluated at T3 time point to observe its relation with LUS scores. LUS refers to "lung ultrasound score" . Accordingly, one hemithorax is divided into 6 zones where the ultrasound probe is placed. If there is only A lines (no consolidation) observed, it is accepted as zero points. If there are three or less B lines (vertical lines that move with the respiration), it refers to 1 point. Four or more vertical B lines refer to 2 points, and lastly distinct visible atelectasis with converged B lines and disrupted pleura refer to 3 points. In total, ultrasonography is applied on 12 different zones, and sum of the points show the actual LUS. Less points mean lungs with better condition, and higher points reflect lungs with atelectasis and consolidation. Therefore a 36 points LUS indicates severely injured lungs.
Intergroup oxygenation difference | Up to 6 hours
  T3 PaO2 values will be compared in laparoscopic and robotic surgery groups.
Perioperative PaCO2 analysis and its relation to T3 LUS | Up to 6 hours
  PaCO2 values will be evaluated at T3 time point to observe its relation with LUS scores. LUS refers to "lung ultrasound score" . Accordingly, one hemithorax is divided into 6 zones where the ultrasound probe is placed. If there is only A lines (no consolidation) observed, it is accepted as zero points. If there are three or less B lines (vertical lines that move with the respiration), it refers to 1 point. Four or more vertical B lines refer to 2 points, and lastly distinct visible atelectasis with converged B lines and disrupted pleura refer to 3 points. In total, ultrasonography is applied on 12 different zones, and sum of the points show the actual LUS. Less points mean lungs with better condition, and higher points reflect lungs with atelectasis and consolidation. Therefore a 36 points LUS indicates severely injured lungs.
Intraoperative compliance change | Up to 6 hours
  dynamic compliance change between T2 and T1.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vuran Yaz I, Bingul ES, Canbaz M, Aygun E, Sanli MO, Ozcan F, Savran Karadeniz M. Evaluation of perioperative lung ultrasound scores in robotic radical prostatectomy: prospective observational study. J Robot Surg. 2025 Mar 11;19(1):112. doi: 10.1007/s11701-025-02272-x. PMID 40069409